CLINICAL TRIAL: NCT03913897
Title: Adiyaman University
Brief Title: The Effect of Virtual Reality and Kaleidoscope on Pain and Anxiety Levels During Venipuncture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2018/5-18
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Pain
Keywords: acute pain; blood collection; nursing; children; distraction
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality group (Experimental): The children in the groups were distracted by virtual reality goggles 2 minutes before venipuncture, until the process was over.
  Interventions: Other: distraction methods
- kaleidoscope group (Experimental): The children in the groups were distracted by kaleidoscope 2 minutes before the blood collection, until the process was over.
  Interventions: Other: distraction methods
- control group (No Intervention): No intervention was made to children in the control group

INTERVENTIONS:
Other: distraction methods — The children in the groups were distracted by virtual reality goggles and kaleidoscope 2 minutes before venipuncture, until the process was over
  Arms: kaleidoscope group; virtual reality group

SUMMARY:
Aim: The study was carried out in randomized control to determine the effect of two different distractions on pain and anxiety during blood collection.

Methods: The population of the study consisted of children between ages of 4-10 years who applied for venipuncture to a training and research hospital in Turkey between July and December 2018. A total of 139 children were included in the study, 46 of them with virtual reality goggles and 43 of them with control group. Information Form, Child Anxiety Scale, Visual Analogue Scale and Wong Baker Pain Scale were used in the collection of data.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 4 and 10 years for the child,
* applying for health control purpose,
* not having any chronic, mental or neurological illness,
* not using any analgesic in the last 6 hours before the venipuncture procedure.

Exclusion Criteria:

-having a chronic, mental or neurological illness,

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Children Fear Scale | 1 minute
  The Children Fear Scale was used to evaluate the children's fear and anxiety. Children Fear Scale is a 0-4 scale, showing five faces that range from a neutral expression (0 = no anxiety) to a frightened face (4 = severe anxiety). Preprocedural and procedural pain, and anxiety were evaluated

SECONDARY OUTCOMES:
Visual Analogue Scale | 1 minute
  The visual analogue scale has been used for evaluating pain levels. Children were asked to mark the level of their pain on a l00 mm., Visual Analogue scale marked at one end as "no pain" and at the other as "worst pain imaginable.
Wong Baker Face Pain Scale | 1 minute
  The Wong Baker Faces scale is a 0-10 scale. Six faces on the cards show a range of emotions from a smiling face (0 very happy/no pain) to a crying face (10 'hurts worst').

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No